CLINICAL TRIAL: NCT05181748
Title: Investigating the Efficiency of Autologous Platelet Rich Plasma Intraovarian Infusion on Improving Ovarian Functionality in Poor Ovarian Response Patients
Brief Title: Autologous Platelet Rich Plasma Intraovarian Infusion for Poor Responders
Acronym: PRPPOR
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genesis Athens Clinic (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenesisAC
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Poor Response to Ovulation Induction; Infertility, Female; Ovarian Insufficiency; Ovarian Failure; Reproductive Sterility; Ovary; Anomaly
Keywords: Autologous platelet rich plasma intraovarian infusion; Assisted reproduction; PRP; In vitro fertilization; Ovarian functionality improvement
MeSH Terms: conditions — Infertility, Female; Infertility; Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: Experimental: Group of participants receiving PRP treatment Women presenting with POR, treated with autologous PRP intraovarian infusion in the mid-luteal phase of the menstrual cycle, undergoing a subsequent stimulated fresh Embryo Transfer-Intracytoplasmic Sperm Injection (ET-ICSI) cycle on the first menstrual cycle following PRP treatment.
  Control Group: Group of participants receiving standard management Women presenting with POR undergoing a stimulated fresh ET-ICSI cycle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Group of participants receiving PRP treatment (Experimental): Women presenting with POR, treated with autologous PRP intraovarian infusion during the mid-luteal phase, undergoing a subsequent stimulated fresh ET-ICSI cycle on the first month following PRP infusion
  Interventions: Biological: Autologous platelet rich plasma
- Control Group: Group of participants receiving standard protocol (No Intervention): Women presenting with POR undergoing a stimulated fresh ET-ICSI cycle

INTERVENTIONS:
Biological: Autologous platelet rich plasma — Preparation of PRP will be performed immediately following blood sample collection. Blood samples will be collected from the median antebrachial vein. PRP will be prepared according to the manufacturer's instructions employing a Regen Autologous Cellular Regeneration (ACR®-C) Kit (Regen Laboratory, Le Mont-sur-Lausanne, Switzerland). Approximately 60 mL of the patient's peripheral blood will be required in order to yield the required volume of PRP. The goal concentration of platelets in PRP is approximately 1.000.000 platelets/µL. The technique of PRP intraovarian infusion resembles the transvaginal paracentesis performed during the oocyte pick-up procedure. Briefly, both ovaries are visualized via transvaginal ultrasound monitoring, and they are intramedullary injected on multiple sites using a 17-gauge single lumen needle, with the patient under inhaled minimal sedation.
  Other Names: PRP
  Arms: Experimental: Group of participants receiving PRP treatment

SUMMARY:
Autologous platelet rich plasma (PRP) intraovarian infusion may improve ovarian response to controlled ovarian stimulation as well as the hormonal profile of poor ovarian response infertile women subjected to intracytoplasmic sperm injection (ICSI) treatment.

DETAILED DESCRIPTION:
Despite recent advances in reproductive medicine, poor ovarian response (POR) management is still considered to be very challenging. Commonly, POR patients present with reduced ovarian reserve and poor ovarian stimulation performance. The POR cycles are characterized by a very limited number of retrieved oocytes, subsequently leading to poor embryo formation and thus to high cycle cancelation rate. Despite the fact that POR constitutes a multifactorial condition, it is well demonstrated that advanced maternal age (AMA) is the most significant contributor of POR. As maternal age increases, reduction of neo-angiogenesis in ovaries is observed, leading to accelerated follicular loss. Considering that PRP contains several growth factors such as vascular endothelial growth factor (VEGF) and cytokines, it has been proposed that intraovarian infusion of autologous PRP could restore the ovarian niche microenvironment, increasing ovarian response to external gonadotropin stimulation. However, limited data are available with regards to PRP efficiency in POR patients, which are mainly originating from pilot or small cohort studies. This interventional non-randomised open-label study aims to investigate the effect of autologous PRP intraovarian infusion on improving POR patient performance by studying a large and well-controlled POR population.

ELIGIBILITY:
Inclusion Criteria:

Poor Ovarian Response according to Bologna Criteria (fulfilling 2 out of 3 of the following):

1. Age ≥ 40 years
2. AMH < 1.1 ng/ml OR AFC < 7
3. ≤ 3 oocytes with a conventional stimulation protocol

   * Discontinuation of any complementary/adjuvant treatment including hormone replacement and acupuncture, for at least three months prior to recruitment.
   * Willing to comply with study requirements

Exclusion Criteria:

* Any pathological disorder related to reproductive system anatomy
* Cycle irregularities
* Amenorrhea
* Endometriosis
* Adenomyosis
* Fibroids and adhesions
* Infections in reproductive system
* Current or previous diagnosis of cancer in reproductive system
* History of familiar cancer in reproductive system
* Severe male factor infertility
* Prior referral for Preimplantation Genetic Testing (PGT) -Ovarian inaccessibility -Endocrinological disorders (Hypothalamus-
* Pituitary disorders, thyroid dysfunction, diabetes mellitus, metabolic syndrome)
* BMI>30 kg/m2 or BMI<18.5 kg/m2
* Systematic autoimmune disorders

Ages: 35 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 34-36 hours following ovulation triggering
  Number of oocytes retrieved following controlled ovarian stimulation in the first fresh ICSI-ET cycle performed on the first menstrual cycle following intervention
Anti-Müllerian Hormone Levels (AMH) | On day 2-3 of the first menstrual cycle post intervention
  Serum anti-müllerian hormone (AMH) levels evaluated in the first menstrual cycle following intervention

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6-7 weeks following last menstruation
  Clinical pregnancy rate, following the first fresh ET-ICSI cycle performed on the first menstrual cycle after intervention
Antral Follicle Count (AFC) | On day 2-3 of the first menstrual cycle post intervention
  Antral Follicle Count (AFC) evaluated in the first menstrual cycle following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Agni Pantou, M.D, Principal Investigator — Genesis Athens Clinic
Locations (1):
- Genesis Athens Clinic, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be provided upon reasonable request, following authorization by the Scientific and Ethical Board of Genesis Athens Clinic